CLINICAL TRIAL: NCT01470144
Title: An Open-label Extension of Study AC-066A301 Investigating the Safety and Tolerability of ACT-385781A in Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: Epoprostenol for Injection in Patients With Pulmonary Arterial Hypertension
Acronym: Epitome2ext
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Collaborators: Chiltern International Ltd. (Industry); Effi-Stat (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-066A302
Record Dates: First submitted 2011-10-28; First posted 2011-11-11 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Epoprostenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Single arm, open-label
  Interventions: Drug: Epoprostenol

INTERVENTIONS:
Drug: Epoprostenol — Administered by continuous intravenous infusion via a central venous catheter; using an ambulatory infusion pump. The dose and infusion rate of EFI may be adjusted throughout the study in order to balance tolerability and maximum clinical benefit

SUMMARY:
This is an open-label, nonrandomized extension to study AC-066A301. The study will assess safety and tolerability of ACT-385781A while providing a means for continuing treatment after ending participation in study AC-066A301.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study-mandated procedure
2. Patients who completed participation in study AC-066A301
3. Patients who have not obtained access for commercial EFI at the time of ending participation in study AC-066A301

Exclusion Criteria:

1. Patients who prematurely discontinued study drug in study AC-066A301
2. Patients for whom continued treatment with EFI is no longer considered appropriate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-07-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Extension study for patients who completed EPITOME-2 (AC-066A301). Patients continued to receive EFI (epoprostenol sodium). In 6 countries (FR, CA, BE, NL, IT, ES) at 8 expert centers for the treatment of patients with pulmonary arterial hypertension. Recruitment started on 15 June 2011 and was completed on 02 February 2012.
Groups:
- Treatment: All patients who received at least one dose of EFI
Period: Overall Study
Arm/Group | Treatment
Started | 41
Completed | 31 ("Completed" corresponds to subjects switching to commercial EFI upon market approval/reimbursement)
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Lung transplant | 6
Not completed — Patient's and investigator's decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: Years] | 46.0 [23 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events
Time Frame: On average 2.72 years
Population: All patients who received at least one dose of EFI
Measure: Number; unit: Number of patients
Arm/Group | Treatment
Number analyzed (Participants) | 41
Number of patients | 41

2. Secondary Outcome: Exposure Duration
Description: Duration of exposure to EFI
Time Frame: On average 2.72 years
Measure: Median (Full Range); unit: year
Arm/Group | Treatment
Number analyzed (Participants) | 41
year | 2.44 [0.5 to 4.0]

ADVERSE EVENTS:
Time Frame: On average 2.72 years
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 35/41
Other Adverse Events (participants affected / at risk) | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=41)
Catheter site infection (Infections and infestations) | 7 (10)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Lung transplant (Surgical and medical procedures) | 6 (6)
Right ventricular failure (Cardiac disorders) | 6 (11)
Device dislocation (General disorders) | 4 (6)
Device related sepsis (Infections and infestations) | 4 (5)
Device occlusion (General disorders) | 3 (3)
Angina pectoris (Cardiac disorders) | 2 (2)
Device alarm issue (General disorders) | 2 (2)
Device damage (General disorders) | 2 (3)
Device leakage (Gastrointestinal disorders) | 2 (2)
Device related infection (Infections and infestations) | 2 (2) — Not local infection, not sepsis
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Transplant evaluation (Investigations) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 1 (1)
Bronchitis moraxella (Infections and infestations) | 1 (1)
Cardiac flutter (Cardiac disorders) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 1 (1)
Catheter site pain (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Device breakage (General disorders) | 1 (1)
Device connection issue (General disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion site vesicles (General disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Medical device change (Surgical and medical procedures) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=41)
Headache (Nervous system disorders) | 12 (15)
Nasopharyngitis (Infections and infestations) | 10 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Diarrhoea (Gastrointestinal disorders) | 10 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Fatigue (General disorders) | 8 (8)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 4 (4)
Bronchitis (Infections and infestations) | 8 (14)
Nausea (Gastrointestinal disorders) | 7 (8)
Palpitations (Cardiac disorders) | 5 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Abdominal distension (Gastrointestinal disorders) | 4 (4)
Gastroenteritis (Infections and infestations) | 4 (5)
Oedema peripheral (General disorders) | 4 (5)
Pyrexia (General disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Catheter site infection (Infections and infestations) | 4 (6)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Asthenia (General disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (4)
Insomnia (Psychiatric disorders) | 3 (3)
Sinusitis (Infections and infestations) | 3 (3)
Weight decreased (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days